CLINICAL TRIAL: NCT05427331
Title: Enterobacteria Capsules in Treatment of Patients With Insomnia Clinical Research on Effectiveness and Safety
Brief Title: FMT Capsules in Treatment of Patients With Insomnia Clinical Research
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yanling Wei, Associate Professor, Department of Gastroenterology, Daping Hospital, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMT-202201
Record Dates: First submitted 2022-06-01; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Chronic Insomnia
Keywords: FMT; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT capsule treatment group (Experimental): drugs use generic name: FMT capsule dosage form: capsule dosage, frequency: 16 capsules once a week duration: 4 weeks
  Interventions: Drug: FMT capsule
- Placebo treatment group (Placebo Comparator): drugs use generic name: Placebo dosage form:capsule dosage,frequency:16 capsules once a week duration:4 weeks
  Interventions: Drug: FMT capsule

INTERVENTIONS:
Drug: FMT capsule — Patients with insomnia need to take FMT capsules orally in an empty stomach in the morning, 16 capsules once a week, for 4 consecutive weeks

SUMMARY:
Objective: To investigate whether Fecal Microbiota Transplantation(FMT) can improve sleep in patients with insomnia, its effect on gut microbiota and its metabolites, and its effect on inflammatory factors, neurotransmitters and sex hormones in peripheral blood. Methods: The study needs to recruit 60 patients with insomnia and randomly divide them into FMT capsule treatment group or Placebo treatment group. The patients were followed up before the treatment and 4, 8, and 12 weeks after the treatment. The sleep status of the patients was assessed by Pittsburgh sleep quality index-PSQI, and the changes of gut microbiota and its metabolites were detected by Metagenomic sequencing and metabonomics analysis.The expression of cytokines, sex hormones and neurotransmitters in peripheral blood were detected by Elisa.

DETAILED DESCRIPTION:
Insomnia is increasingly common in modern society. In recent years, more and more studies have shown that compared with healthy people, insomnia patients have changes in gut microbiota and its metabolites. At the same time, gut microbiota, as an important part of the gastrointestinal tract, can affect the stability of the body's internal environment through a variety of ways through the "microbial-gut-brain axis", including the regulation of immune response. However, relevant studies at home and abroad mainly focus on sleep deprivation, while there are few reports on the intervention of gut microbiota in insomnia. The purpose of this study was to investigate whether Fecal Microbiota Transplantation(FMT) can improve sleep in patients with insomnia, its effect on gut microbiota and its metabolites,and its effect on inflammatory factors, neurotransmitters and sex hormones in peripheral blood. The study needs to recruit 60 patients with insomnia and randomly divide them into FMT capsule treatment group or Placebo treatment group. The patients were followed up before the treatment and 4, 8, and 12 weeks after the treatment. The sleep status of the patients was assessed by Pittsburgh sleep quality index-PSQI, and the changes of gut microbiota and its metabolites were detected by Metagenomic sequencing and metabonomics analysis.The expression of cytokines, sex hormones and neurotransmitters in peripheral blood were detected by Elisa.

ELIGIBILITY:
Inclusion Criteria:

* 1) Men and women are not limited, the age is 18-70 years old; 2) The course of disease is more than 3 months, and the diagnosis is insomnia (refer to the diagnostic criteria of insomnia in the International Classification of Sleep Disorders Third Edition (ICSD3), and Pittsburgh sleep quality index-PSQI>15 points); 3) The vital signs are stable, the consciousness is clear, there is no communication and cognitive impairment, and can cooperate with the questionnaire; 4) Agree to participate in the research and sign the informed consent; 5) Able to receive follow-up examinations, follow-up examinations and collection of specimens on time.

Exclusion Criteria:

* 1) The patients took probiotics or prebiotics products within 3 months before the research; 2) The patient took antibiotics within 3 months before the research; 3) The patient smokes heavily (≥10 cigarettes/day), or is dependent on alcohol, coffee, or strong tea; 4) The Patients rely on tube feeding; 5) The patient has a history of severe allergies; 6) The patient has severe organic disease; 7) The patient cannot cooperate to complete the study; 8) Pregnant or lactating women; 9) The patient has depression, anxiety, schizophrenia or other serious mental illness; 10) The Patients with insomnia due to physical diseases or mental disorders; 11) Other patients deemed unsuitable for inclusion by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
PSQI scale was used to assess sleep | FMT capsule/placebo treatment after 4 weeks
  Pittsburgh sleep quality index scale was used to assess sleep

SECONDARY OUTCOMES:
The metagenomic measure the types of gut microbiota | FMT capsule/placebo treatment after 4 weeks
  The metagenomic measure the types of gut microbiota

OTHER OUTCOMES:
The concentration of serotonin | FMT capsule/placebo treatment after 4 weeks
  The concentration of serotonin by ELISA
The concentration of norepinephrine | FMT capsule/placebo treatment after 4 weeks
  The concentration of norepinephrine by ELISA
The concentration of dopamine | FMT capsule/placebo treatment after 4 weeks
  The concentration of dopamine by ELISA
The concentration of ϒ- aminobutyric acid | FMT capsule/placebo treatment after 4 weeks
  The concentration of ϒ- aminobutyric acid by ELISA
The concentration of melatonin | FMT capsule/placebo treatment after 4 weeks
  The concentration of melatonin by ELISA
The concentration of interleukin-6 | FMT capsule/placebo treatment after 4 weeks
  The concentration of interleukin-6 by ELISA
The concentration of interleukin-1 β | FMT capsule/placebo treatment after 4 weeks
  The concentration of interleukin-1 β by ELISA
The concentration of tumor Necrosis Factor -α | FMT capsule/placebo treatment after 4 weeks
  The concentration of tumor Necrosis Factor -α by ELISA
The concentration of interleukin-10 | FMT capsule/placebo treatment after 4 weeks
  The concentration of interleukin-10 by ELISA
The concentration of follicle-stimulating hormone | FMT capsule/placebo treatment after 4 weeks
  The concentration of follicle-stimulating hormone by ELISA
The concentration of estradiol | FMT capsule/placebo treatment after 4 weeks
  The concentration of estradiol by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Yanling Wei, Study Director — Third Military Medical University
Locations (1):
- Third Military Medical University Daping Hospital, Chongqing, Chongqing Municipality, China